CLINICAL TRIAL: NCT06110468
Title: Tailored Follow-up for Persons With Multiple Sclerosis to Optimize Physical Functions, Health and Employment: a Prospective Single-blinded Randomized Controlled Trial
Brief Title: Physical Function, Health and Employment for People With Multiple Sclerosis
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nordlandssykehuset HF (Other)
Collaborators: The Royal Norwegian Ministry of Health (Other); University Hospital of North Norway (Other); Nord University (Other); UiT The Arctic University of Norway (Other); Helgeland Hospital Trust (Other); University of Tasmania (Other); Norwegian Labour and Welfare Administration (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: HNF1687-23
Record Dates: First submitted 2023-10-24; First posted 2023-10-31 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Multiple Sclerosis
Keywords: Physiotherapy; Employment; Physical activity; Health related quality of life; Cost-benefit
MeSH Terms: conditions — Multiple Sclerosis; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention, CoreDISTParticpation (Experimental): Week 1-2: a)Videos for PwMS and employers on MS, possible work adaptations, physical activity (PA) and function. b)A meeting between PwMS and a work-consultant (WC). They will decide if the PwMS should discuss the work situation with their employer or if the WC and/or other professionals are needed. c)A clinical assessment with a trained MS-OP-PT to explore possibilities for optimalisation of movement.
  Week 3-8: a)A clinical assessment with the mPT building on previous assessment. Goal-setting for function and PA. b)CoreDIST-training in groups, 6 weeks, 1/week. indoors and 1/week outdoors. Independent training 1/week, CoreDISTvideos. c)A follow up meeting regarding work, evaluation of goals with mPT. New goal setting for week 10-15 Week 10-15, Self-administered, digitally supported home training: a)CoreDIST-videos 3x10 min/week b)Training of own choice including elements of high intensity and balance 2x30 minutes per week. c)Week 15: Evaluation of goals regarding work and PA
  Interventions: Other: CoreDISTParticipation
- Control, usual care (No Intervention): Usual care (control group): These participants will continue with their regular routines and will be encouraged to obtain the national and MS-specific recommendation of 150-300 minutes of moderate physical activity or 75 minutes of high intensity physical activity per week or a combination of these, stay employed, continue medical treatment and seek any health care required, including physiotherapy.

INTERVENTIONS:
Other: CoreDISTParticipation — CoreDISTparticipation is a multi-disciplinary individualized intervention that concurrently combine 1) providing PwMS and their employers with information on MS, possibilities for work-adaptations within the welfare system and the importance of physical activity 2) Structured goal-setting regarding reducing barriers for work and regarding physical function and activity for PwMS 3) A physiotherapy intervention focusing on improving the underlying prerequisites for balance and walking along with high intensive training and promotion of physical activity 4) structured evaluation and adjustment of goals.
  Arms: Intervention, CoreDISTParticpation

SUMMARY:
Employment is low in people with MS, even when physical levels of functioning are high. The purpose of this study is to investigate if an individually tailored intervention combining individualized physiotherapy and work adaptation works better than usual care in terms of reducing barriers for work and improving levels of physical activity. The utility of the intervention will be investigated in terms of quality adjusted life years, long-term employment status and work-related costs.

DETAILED DESCRIPTION:
Physiotherapy and physical activity interventions can reduce fatigue, improve balance, walking, HRQoL, and may improve neuromuscular and physical functioning in people with MS. However, these interventions lack coordination between health care levels and sectors and rarely address vital employment adaptations. Optimizing function and physical activity, when disability is low and neuroplasticity is optimal, can be valuable for maintaining work as levels of fatigue, mobility related symptoms and cognitive disturbances are associated with current employment.

People with an MS-diagnosis who reside in the North of Norway will be identified from patient lists from the neurological out-patient clinics in the participating hospitals. Upon the provision of written informed consent, all participants will undergo baseline testing prior to randomization into either the intervention or the control group. The intervention group will receive a physiotherapy assessment at the hospitals focusing on opportunities for change. Following this assessment they will participate in group training with a municipality physiotherapist twice weekly for six weeks followed by independent training for six weeks. In addition, both participants and their employers will get access to information films on opportunities for work adaptations and the importance of physical activity. Structured meetings with a specially trained employment consultant, the participant and their employer will be held to discuss possible work adaptations. Goals will be set and formally evaluated. Retests will be carried out at week 9, 16 and 52. Registry data on employment will be obtained from the Norwegian labour and welfare administration as a part of a cost-benefit analysis of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Multiple Sclerosis according to the McDonald's criteria
* Extended Disability Status Scale (EDSS) 0-4
* Being employed, part time or full time, may include various degrees of sick leave, disability pension or AAP.
* Living in the participating 18 municipalities (Hammerfest, Alta, Senja, Målselv, Tromsø, Harstad, Narvik, Fauske, Bodø, Meløy, Vågan, Vestvågøy, Sortland, Hadsel, Rana, Vefsn, Alstadhaug, Brønnøy).

Exclusion Criteria:

* Pregnancy at enrolment.
* Exacerbation of symptoms (i.e. relapse) within two weeks prior to enrolment.
* Other serious conditions.

Ages: 18 Years to 67 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Estimated)
Dates: Start 2024-03-04 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2035-12 (Estimated)

PRIMARY OUTCOMES:
Multiple Sclerosis Work Difficulties Questionnaire -23 Norwegian version | Baseline, 9, 16 and 52 weeks post baseline
  How frequently individuals with MS perceive psychological/cognitive (11 items), physical (8 items), external, (4 items) barriers related to work, scored by a 5-point scale (0=best).
Levels of physical activity measured using ActiGraph wGT3x-BT monitors | Participants will wear device for one week after testing at baseline and at 9, 16 and 52 weeks post baseline
  % of time in mild, moderate, intensive physical activity and sedate time

SECONDARY OUTCOMES:
6 meter walk test | Baseline, 9, 16 and 52 weeks post baseline
  Walking distance (meters) within six minutes
Step count using ActiGraph wGT3x-BT monitors | Participants will wear device for one week after testing at baseline and at 9, 16 and 52 weeks post baseline
  Daily average number of steps
Fatigue Severity Scale -Norwegian version | Baseline, 9, 16 and 52 weeks post baseline
  Self-report, 9 items: physical, social and cognitive effects of fatigue, scale:1-7 (high score indicates higher levels of fatigue).
Multiple Sclerosis Walking Scale-12 | Baseline, 9, 16 and 52 weeks post baseline
  Self-reported perception of walking, 12 items, score on a 5-point scale. Higher score indicate higher impact of MS on the individuals walking ability.
Mini Balance Evaluation Systems Test (MiniBESTest) | Baseline, 9, 16 and 52 weeks post baseline
  Pro-and reactive balance, dual task and involving sit to stand, standing and walking, 14 items on a 3-point scale. Higher score indicate better performance.
Trunk Impairment Scale-modified Norwegian version (TISmodNV) | Baseline, 9, 16 and 52 weeks post baseline
  Trunk control in sitting. 6 items, score on a 2- or 3-point scale, sum range 0-16 points. Higher score indicates higher levels of trunk control.
Postural control measured by AccuGait Optimized force platforms | Baseline, 9, 16 and 52 weeks post baseline
  Measures postural control in standing, tandem, one-leg standing: postural sway of center of pressure.
European Quality of Life 5-Dimension (EQ-5D-5L) + Complementary questions | Baseline, 9, 16 and 52 weeks post baseline
  Self-perceived HRQoL regarding five domains, and a VAS scale (0-100) on overall health.
  Complementary questions on sleep, wellbeing, emotions, social relations (advocated by the Norwegian Health Institute). Higher score indicate better self-perveived health.
Multiple Sclerosis Impact Scale 29-Norwegian version | Baseline, 9, 16 and 52 weeks post baseline
  Self-perceived physical (13 items), psychological (9 items) impact on HRQoL, a 5-point scale. Higher score indicate increased impact of MS on the individuals day-to-day life.
Patient Global Impression of Change - physical activity and balance | Baseline, 9, 16 and 52 weeks post baseline
  A global index that is used to rate the response of a condition to a therapy (transition scale). Higher score indicate improvement.

CONTACTS AND LOCATIONS:
Locations (1):
- Nordlandssykehuset HF, Bodø, Nordland, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Normann B, Sivertsen M, Braaten TB, Melberg HO, Fikke HK, Elvik M, Arntzen EC. A Comprehensive and Structured Follow-Up for Persons With Multiple Sclerosis (CoreDISTparticipation) to Optimize Physical Functions, Health, and Employment: Protocol for a Prospective, Single-Blinded Randomized Controlled Trial and Health Economic Evaluation. JMIR Res Protoc. 2025 Oct 8;14:e74988. doi: 10.2196/74988. PMID 41061251